CLINICAL TRIAL: NCT06704893
Title: The Efficacy of Amniotic Suspension Allograft Injection in the Treatment of Knee Osteoarthritis: a Randomized Double-blind Controlled Trial
Brief Title: Amniotic Suspension Allograft Injection for Knee Osteoarthritis
Acronym: ASAIKO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Po-Cheng Chen, Assistant professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202401278A3
Record Dates: First submitted 2024-10-26; First posted 2024-11-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Knee; Osteoarthritis
Keywords: double-blind randomized controlled trial; amniotic suspension allograft injection; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (4):
- ASA injection 40 mg group (Experimental): AMNIOGEN® 40mg (HCT Regenerative, New Taipei, Taiwan) was diluted in 3.0 mL of sterile normal saline.
  Interventions: Drug: ASA injection 40 mg group
- ASA injection 20 mg group (Experimental): AMNIOGEN® 20mg (HCT Regenerative, New Taipei, Taiwan) was diluted in 3.0 mL of sterile normal saline.
  Interventions: Drug: ASA injection 20 mg group
- HA injection group (Active Comparator): 3 ml of HyLink (SEIKAGAKU CORPORATION, Tokyo, Japan)
  Interventions: Drug: HA injection group
- Normal saline injection group (Placebo Comparator): 3 ml of sterile normal saline
  Interventions: Drug: Normal saline injection group

INTERVENTIONS:
Drug: ASA injection 40 mg group — Participants will receive intra-articular knee injections under ultrasound guidance with AMNIOGEN® 40mg (HCT Regenerative, New Taipei, Taiwan) diluted in 3.0 mL of sterile normal saline.
  Arms: ASA injection 40 mg group
Drug: ASA injection 20 mg group — Participants will receive intra-articular knee injections under ultrasound guidance with AMNIOGEN® 20mg (HCT Regenerative, New Taipei, Taiwan) diluted in 3.0 mL of sterile normal saline.
  Arms: ASA injection 20 mg group
Drug: HA injection group — Participants will receive intra-articular knee injections under ultrasound guidance with 3 ml of HyLink (SEIKAGAKU CORPORATION, Tokyo, Japan).
  Arms: HA injection group
Drug: Normal saline injection group — Participants will receive intra-articular knee injections under ultrasound guidance with 3 ml of sterile normal saline.
  Arms: Normal saline injection group

SUMMARY:
There have been few clinical trials on ASA for the treatment of knee osteoarthritis, and there is currently no literature reporting the optimal treatment dosage. Non-surgical treatment options include braces, weight loss, lifestyle changes, oral pain relievers, and intra-articular injections. Recently, placental-derived tissues have gradually been applied in the treatment of knee osteoarthritis. These tissues were initially used primarily for burns, ulcers, and wounds that are difficult to heal, but have now begun to be utilized in the orthopedic field. They have been proven to contain various anti-inflammatory cytokines and growth factors, which can reduce inflammation associated with arthritis. Reducing inflammation not only alleviates the pain of knee osteoarthritis but also improves patients' quality of life. The purpose of this study is to compare the therapeutic effects of amniotic suspension allograft (ASA), hyaluronic acid (HA), and saline on knee osteoarthritis and to examine whether there is a dose-response relationship with ASA injections.

DETAILED DESCRIPTION:
According to statistics from the Ministry of Health and Welfare, the prevalence of knee osteoarthritis in Taiwan is approximately 15%. The main causes of the disease include overuse of joint cartilage and abnormal synovial fluid secretion, which impair joint mobility and cause symptoms like pain, swelling, and warmth. In severe cases, bone spurs and joint deformities can develop, further limiting mobility. Non-surgical treatment options for knee osteoarthritis currently include the use of braces, weight loss, lifestyle changes, oral pain relievers, and intra-articular injections, with only a small number of patients requiring surgery due to severe joint cartilage wear. In terms of injection treatments, given the limited efficacy of traditional corticosteroid and HA injections for knee osteoarthritis, an increasing number of physicians are using platelet-rich plasma (PRP) injections. Numerous clinical trials have supported this treatment option. However, the effectiveness of PRP treatment is partly dependent on the quality of the patient's blood. If the patient has poor blood quality (e.g., due to old age, multiple chronic diseases, autoimmune disorders, or use of anticoagulants), the efficacy of PRP injections will be significantly reduced.

Recently, a highly promising treatment option-placental-derived tissues-has begun to be used for knee osteoarthritis. Historically, placental-derived tissues have been applied to burns, ulcers, and other difficult-to-heal wounds such as corneal ulcers. More recently, these tissues have been applied in the orthopedic field. These products come in several formulations, some containing pulverized tissues (amniotic membrane, chorion, or both), cells from amniotic fluid, amniotic fluid itself, or a combination of these components. Placental tissues have been shown to contain a variety of anti-inflammatory cytokines, growth factors, and inhibitors, which are believed to reduce the inflammatory response associated with arthritis. Reducing this inflammation can not only alleviate the pain of knee osteoarthritis but also improve the quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Body mass index (BMI) less than 40 kg/m².
3. Symptomatic knee osteoarthritis with X-ray evidence graded 2 or 3 on the Kellgren-Lawrence (KL) grading scale.
4. Numerical Rating Scale (NRS) score (scale 1 to 10) for pain greater than 4 over the past 7 days.
5. Able to walk independently or with the aid of a cane.

Exclusion Criteria:

1. Pregnant women or women planning pregnancy.
2. Regular use of anticoagulants.
3. Use of pain medications (except acetaminophen) within 15 days prior to injection.
4. History of substance abuse.
5. Patients who take additional knee symptom-relief medications during the study must report it to the research team; failure to comply will result in exclusion.
6. Corticosteroid or visco-supplementation injection into the affected knee within 3 months prior to enrollment.
7. Knee surgery on the affected side within 12 months before enrollment, or surgery on the contralateral knee within 6 months before enrollment.

9. History of organ or hematopoietic stem cell transplant. 11. Current use of immunosuppressive agents. 12. Diagnosis of cancer within the past 5 years (except for treated basal cell carcinoma).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | From enrollment to the end of study at 12 months
  This scale assesses overall pain severity, with scores ranging from 0 (no pain) to 10 (severe pain). Measurements will be taken before treatment and at 1, 3, 6, and 12 months after treatment.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | From enrollment to the end of study at 12 months
  This questionnaire measures knee injury and osteoarthritis impact across five domains: pain, symptoms, activities of daily living (ADL), sport and recreation function, and quality of life. Measurements will be collected at baseline and at 1, 3, 6, and 12 months post-treatment. The resulting scores are transformed to a scale from 0 (extreme knee problems) to 100 (no knee problems).
The World Health Organization Quality of Life Brief Version (WHOQOL-BREF) | From enrollment to the end of study at 12 months
  This quality-of-life assessment, developed by the World Health Organization, evaluates four domains: physical health, psychological well-being, social relationships, and environment. It will be administered before treatment and at 1, 3, 6, and 12 months post-treatment. The score of each domain ranges from 0 (worst outcome) to 100 (best outcome). The total score is the summation of each domain score.

SECONDARY OUTCOMES:
Number of participants with abnormal Complete Blood Count (CBC) | From enrollment to the end of study at 12 months
  Each participant will undergo blood tests for Complete Blood Count (CBC) before treatment, and at 1 month, 3 months, 6 months, and 12 months after treatment. Complete Blood Count (CBC) includes
  1. WBC in 1000/μL
  2. RBC in million/μL
  3. Hemoglobin in g/dL
  4. Hematocrit in %
  5. MCV in fL
  6. MCH in pg/cell
  7. MCHC in g/dL
  8. RDW in %
  9. RDW-SD in fL
  10. Platelet in 1000/μL
  11. PDW in fL
  12. MPV in fL All blood samples will be analyzed at the laboratory of Chang Gung Memorial Hospital. The investigators will count the number of participants with abnormal CBC.
C-reactive protein (CRP) | From enrollment to the end of study at 12 months
  Each participant will undergo blood test for C-reactive protein (CRP in mg/L) before treatment, and at 1 month, 3 months, 6 months, and 12 months after treatment. All blood samples will be analyzed at the laboratory of Chang Gung Memorial Hospital.
Erythrocyte Sedimentation Rate (ESR) | From enrollment to the end of study at 12 months
  Each participant will undergo blood test for Erythrocyte Sedimentation Rate (ESR in mm/hr) before treatment, and at 1 month, 3 months, 6 months, and 12 months after treatment. All blood samples will be analyzed at the laboratory of Chang Gung Memorial Hospital.
Cytokine IL-6 | From enrollment to the end of study at 12 months
  Each participant will undergo blood test for cytokine IL-6 in pg/mL before treatment, and at 1 month, 3 months, 6 months, and 12 months after treatment. All blood samples will be analyzed at the laboratory of Chang Gung Memorial Hospital.
Knee Ultrasound Imaging | From enrollment to the end of study at 12 months
  Each participant will undergo ultrasound evaluation before treatment, and at 1 month, 3 months, 6 months, and 12 months after treatment. The evaluation will mainly assess the volume of effusion, the degree of damage to the medial and lateral femoral trochlear cartilage17 (grade 0: normal; grade 1: slightly blurred cartilage edges or increased echogenicity of the cartilage; grade 2A: partial thinning of the cartilage, thinning <50% of the original cartilage thickness; grade 2B: partial thinning of the cartilage, thinning >50% of the original cartilage thickness; grade 3: complete loss of cartilage thickness), and whether there is meniscus extrusion in the medial or lateral meniscus.
Knee X-ray | From enrollment to the end of study at 12 months
  Each participant will undergo knee X-rays (AP view, lateral view, merchant view) at baseline and 12 months post-treatment.
Cartilage Oligomeric Matrix Protein (COMP) | From enrollment to the end of study at 12 months
  Each participant will undergo blood test for Cartilage Oligomeric Matrix Protein (COMP in IU) before treatment, and at 1 month, 3 months, 6 months, and 12 months after treatment. All blood samples will be analyzed at the laboratory of Chang Gung Memorial Hospital.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung, Taiwan
  - Department of Physical Medicine and Rehabilitation, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City

IPD SHARING:
Plan to Share IPD: Undecided
Secondary analysis might be performed after the primary study, so IPD will not be shared immediately after finishing the study